CLINICAL TRIAL: NCT04048512
Title: Circulating Tumor Cells (CTC) Before and After Thoracic Resection With and Without Intraoperative Use of Extra Coprporeal Membrane Oxygenator (ECMO) or Cardio Pulmonary By Pass (CPB)
Brief Title: Circulating Tumor Cells (CTC) Before and After Thoracic Resection With and Without Intraoperative Use of ExtraCorporeal Membrane Oxygenator(ECMO) or Cardio Pulmonary By Pass (CPB)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: R1005/19-IEO 1060
Record Dates: First submitted 2019-08-02; First posted 2019-08-07 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Thoracic Surgery; Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Resection with intraoperative ECMO/CPB: Patients suffering of neoplastic thoracic disease, undergoing thoracic resection with intraoperative use of Extra Corporeal Membrane Oxygenator (ECMO) or Cardio Pulmonary By pass (CPB)
  Interventions: Procedure: Resection with intraoperative use of ECMO/CPB
- Resection without intraoperative ECMO/CPB: Patients suffering of neoplastic thoracic disease, undergoing thoracic resection without intraoperative use of Extra Corporeal Membrane Oxygenator (ECMO) or Cardio pulmonary By Pass (CPB)
  Interventions: Procedure: Resection without intraoperative use of ECMO/CPB

INTERVENTIONS:
Procedure: Resection with intraoperative use of ECMO/CPB — Patients are operated with the use of intraoperative ECMO/CPB
  Groups: Resection with intraoperative ECMO/CPB
Procedure: Resection without intraoperative use of ECMO/CPB — Patients are operated without the use of intraoperative ECMO/CPB
  Groups: Resection without intraoperative ECMO/CPB

SUMMARY:
The role of circulating tumor cells (CTC) in patients suffering from lung cancer and thoracic malignancies is not well known and it is still widely debated. The use of intraoperative cardiorespiratory supports like ECMO (extracorporeal membrane oxygenator) and CPB (cardiopulmonary by-pass) during extended resections in oncologic patients has been questioned because of the theoretical risk of tumor cells spreading, although there is no clinical or experimental evidence supporting this hypothesis.

The aim of the present study is to quantify the possible presence and amount of CTC in the peripheral blood of patients undergoing lung/mediastinal resection, before and after surgical procedure, comparing patients receiving intraoperative cardiorespiratory support with patients - with similar oncologic disease and extension - operated without the need of ECMO or CPB.

DETAILED DESCRIPTION:
Background and Rationale:

Locally advanced pulmonary and mediastinal cancers invading vital structure such as heart, great vessels, or carina cancer are generally considered as unresectable and incurable. Complete resection in healthy tissue may be compromised due to the proximity of the tumors to vital organs [1, 2]. Palliation with chemotherapy and/or radiotherapy is the principal means of treatment [1, 2]. In highly selected patients with specific anatomic conditions, complete R0 resection for locally advanced tumor has been reported with prolonged survival and, on occasion, resulted in cure [3-5]. Complex cardiac resections or reconstructions, replacement of the thoracic aorta, or the common pulmonary artery can only be approached with cardiac arrest and total circulatory support by standard cardio-pulmonary bypass (CPB) [6,7]; extracorporeal membrane oxygenation (ECMO) is a well- established technique for the management of respiratory or hemodynamic disturbance during lung transplantation. Technological advances in pumps, cannulae, and oxygenators and growing experience for thoracic surgeon during lung transplantation have led to the use of ECMO during conventional thoracic surgical procedure [8,9].

A theoretical possibility of enhancement of metastasis due to ECMO or CPB has been reported [10] although no clear evidence exists ; nevertheless, due to the lack of data about this aspect, many cardio-thoracic surgeons are skeptical about the use of intraoperative CPB or ECMO .

The aim of this protocol is to assess the presence or not and possibly the amount of CTC before and after surgery in the peripheral blood of patients undergoing thoracic resection with (experimental arm) or without (control arm) intraoperative support of ECMO or CPB.

Study design and duration Prospective, double arm , observational study.

Ten consecutive patients - with thoracic malignancies undergoing resection with planned intraoperative cardiorespiratory support - will be enrolled. Before surgery peripheral blood samples will be collected (as subsequently described) to search the presence and the amount of CTC. The patients will then undergo surgical procedure with intraoperative ECMO or CPB support. After the procedure peripheral blood samples will be collected as previously reported to search for CTC.

Ten consecutive patients, presenting the same neoplastic diseases of the experimental arm and with same extension but not requiring intraoperative ECMO or CPB support will be enrolled in the control arm, receiving the same blood sample collection before and after surgery, to assess the presence and the amount of CTC.

The two groups will be than compared in terms of preoperative and postoperative CTC presence and amount.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic resection (lung and or mediastinal resection) requiring intraoperative Extra Coprporeal Membrane Oxygenator (ECMO) or Cardio Pulmonary By pass (CPB) support; in the control group same disease and planned procedure to be performed without the need of EMCO or CPB.
* Infiltration of the main carina
* Infiltration of superior vena cava
* Single lung surgery
* Mediastinal involvment

Exclusion Criteria:

* Age younger than 18 years
* Contraindications to general anesthesia
* Poor general clinical conditions ( ECOG PS >=2)
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ten consecutive patients with planned intraoperative cardiorespiratory support will be enrolled and blood samples will be collected to search for CTC. The patients will then undergo operation with Extra Corporeal membarne Oxygenator (ECMO) or Cardio Pulmonary By Pass (CPB) support. After the procedure peripheral blood samples will be collected as previously reported to search for Circulating Tumor Cells (CTC).
  Ten consecutive patients, presenting the same neoplastic diseases of the experimental arm and with same extension but not requiring intraoperative ECMO or CPB support will be enrolled in the control arm, receiving the same blood sample collection before and after surgery, to assess the presence and the amount of CTC.
  The two groups will be than compared in terms of preoperative and postoperative CTC presence and amount.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the number of circulating tumor cells the day before surgery and first post operative day (24 hours after surgery) | The day before surgery and the first post operative day (24 hours after surgery)
  Quantification of CTC (number) in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Petrella, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institue of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spira A, Ettinger DS. Multidisciplinary management of lung cancer. N Engl J Med. 2004 Jan 22;350(4):379-92. doi: 10.1056/NEJMra035536. No abstract available. PMID 14736930
- [Background] Rice TW, Blackstone EH. Radical resections for T4 lung cancer. Surg Clin North Am. 2002 Jun;82(3):573-87. doi: 10.1016/s0039-6109(02)00017-8. PMID 12371586
- [Background] Regnard JF, Perrotin C, Giovannetti R, Schussler O, Petino A, Spaggiari L, Alifano M, Magdeleinat P. Resection for tumors with carinal involvement: technical aspects, results, and prognostic factors. Ann Thorac Surg. 2005 Nov;80(5):1841-6. doi: 10.1016/j.athoracsur.2005.04.032. PMID 16242466
- [Background] de Perrot M, Fadel E, Mercier O, Mussot S, Chapelier A, Dartevelle P. Long-term results after carinal resection for carcinoma: does the benefit warrant the risk? J Thorac Cardiovasc Surg. 2006 Jan;131(1):81-9. doi: 10.1016/j.jtcvs.2005.07.062. Epub 2005 Dec 5. PMID 16399298
- [Background] Perentes J, Bopp S, Krueger T, Gonzalez M, Jayet PY, Lovis A, Matzinger O, Ruffieux C, Ris HB, Letovanec I, Peters S. Impact of lung function changes after induction radiochemotherapy on resected T4 non-small cell lung cancer outcome. Ann Thorac Surg. 2012 Dec;94(6):1815-22. doi: 10.1016/j.athoracsur.2012.08.054. Epub 2012 Oct 25. PMID 23103000
- [Background] Tsuchiya R, Asamura H, Kondo H, Goya T, Naruke T. Extended resection of the left atrium, great vessels, or both for lung cancer. Ann Thorac Surg. 1994 Apr;57(4):960-5. doi: 10.1016/0003-4975(94)90214-3. PMID 8166550
- [Background] Rao V, Todd TR, Weisel RD, Komeda M, Cohen G, Ikonomidis JS, Christakis GT. Results of combined pulmonary resection and cardiac operation. Ann Thorac Surg. 1996 Aug;62(2):342-6; discussion 346-7. PMID 8694588
- [Background] Lang G, Ghanim B, Hotzenecker K, Klikovits T, Matilla JR, Aigner C, Taghavi S, Klepetko W. Extracorporeal membrane oxygenation support for complex tracheo-bronchial proceduresdagger. Eur J Cardiothorac Surg. 2015 Feb;47(2):250-5; discussion 256. doi: 10.1093/ejcts/ezu162. Epub 2014 Apr 16. PMID 24740936
- [Background] Lang G, Taghavi S, Aigner C, Charchian R, Matilla JR, Sano A, Klepetko W. Extracorporeal membrane oxygenation support for resection of locally advanced thoracic tumors. Ann Thorac Surg. 2011 Jul;92(1):264-70. doi: 10.1016/j.athoracsur.2011.04.001. PMID 21718853
- [Background] Brutel de la Riviere A, Knaepen P, Van Swieten H, Vanderschueren R, Ernst J, Van den Bosch J. Concomitant open heart surgery and pulmonary resection for lung cancer. Eur J Cardiothorac Surg. 1995;9(6):310-3; discussion 313-4. doi: 10.1016/s1010-7940(05)80188-5. PMID 7546803